CLINICAL TRIAL: NCT05997238
Title: Evaluation of the Effect of Triamcinolone at Different Doses on Local Infiltration Anesthesia During Total Knee Arthroplasty
Brief Title: Evaluation of the Effect of Triamcinolone at Different Doses on LIA During TKA
Acronym: LIA;TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Triamcinolone68480
Record Dates: First submitted 2023-05-17; First posted 2023-08-18 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2023-04

CONDITIONS: Osteoarthritis, Knee
Keywords: total knee arthroplasty; triamcinolone; local infiltration anesthesia
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Triamcinolone

STUDY DESIGN:
Intervention Model Description: An independent researcher, who would not meet or interact with patients before recruiting them, compiled a computer-generated randomised list using a 1:1:1:1 assignment and random blocks of 12, 8 or 4 to ensure the concealability of the assignment. The groups corresponding to the numbers generated by the random number generator were placed in opaque envelopes and sealed, and the enrolled patients were assigned envelopes in the chronological order in which they were enrolled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent researcher, who would not meet or interact with patients before recruiting them, compiled a computer-generated randomised list using 1:1 assignments and random blocks of 8, 6 or 4 to ensure the invisibility of assignments. The groups corresponding to the numbers generated by the random number generator were placed in opaque envelopes and sealed, and the enrolled patients were assigned envelopes in the chronological order in which they were enrolled. On the day of surgery, the anesthesiologist prepares to mix the drug preparation after opening the sealed envelope, which is then handed to the operating room nurse. The patient, the rehabilitation physician, and the ward nurse did not know the type of drug mixture the patient was injected with.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): LIA preparation was administered without triamcinolone. The base formula contains 150mg ropivacaine and 0.5mg epinephrine. Add normal saline and mix to 80ml.
  Interventions: Drug: without triamcinolone
- Low dose triamcinolone (Experimental): Add 20mg triamcinolone to the LIA preparation. The base formula contains 150mg ropivacaine and 0.5mg epinephrine. Add normal saline and mix to 80ml.
  Interventions: Drug: 20mg triamcinolone
- Moderate dose triamcinolone (Experimental): add 40mg triamcinolone to the LIA preparation. The base formula contains 150mg ropivacaine and 0.5mg epinephrine. Add normal saline and mix to 80ml.
  Interventions: Drug: 40mg triamcinolone
- High dose triamcinolone (Experimental): add 80mg triamcinolone to the LIA preparation. The base formula contains 150mg ropivacaine and 0.5mg epinephrine. Add normal saline and mix to 80ml.
  Interventions: Drug: 80mg triamcinolone

INTERVENTIONS:
Drug: without triamcinolone — The preparation contains only the basic formula. The base formula contains 150mg ropivacaine and 0.5mg epinephrine. Add normal saline and mix to 80ml.
  Other Names: Placebo
  Arms: Placebo
Drug: 20mg triamcinolone — 20mg triamcinolone was added to the preparation. Mix 20mg triamcinolone and the basic formula to make a mixed preparation. The base formula contains 150mg ropivacaine and 0.5mg epinephrine. Add normal saline and mix to 80ml.
  Other Names: Low dose triamcinolone
  Arms: Low dose triamcinolone
Drug: 40mg triamcinolone — 40mg triamcinolone was added to the preparation. Mix 40mg triamcinolone and the basic formula to make a mixed preparation. The base formula contains 150mg ropivacaine and 0.5mg epinephrine. Add normal saline and mix to 80ml.
  Other Names: Moderate dose triamcinolone
  Arms: Moderate dose triamcinolone
Drug: 80mg triamcinolone — 80mg triamcinolone was added to the preparation. Mix 80mg triamcinolone and the basic formula to make a mixed preparation. The base formula contains 150mg ropivacaine and 0.5mg epinephrine. Add normal saline and mix to 80ml.
  Other Names: High dose triamcinolone
  Arms: High dose triamcinolone

SUMMARY:
To evaluate the efficacy and safety of different doses of triamcinolone for local infiltration analgesia during total knee replacement

DETAILED DESCRIPTION:
Participants were enrolled according to protocol requirements. Patients who meet all inclusion criteria and do not have any exclusion criteria will be considered for inclusion in the study and will provide the relevant information used orally and in writing. Patients were divided into four groups according to the dose of triamcinolone in the peripheral infiltrating anesthetic preparation. All of which are appropriate for their surgical treatment, and the purpose of the study is to determine which formula is clinically better. All patients enrolled in this study were voluntary participants and signed informed consent. On the day of the surgery, the anesthesiologist prepares a mixture of medications based on patient groups, which are then handed to the operating room nurse. The timing, dose, and site of injection were consistent. Before the prosthesis is installed, the mixture is injected into the upper part of the patella, the posterior joint capsule, and the patellar tendon. After the prosthesis was installed, the mixture was injected into the lateral joint capsule and subcutaneous tissue. The patient, the rehabilitation physician, and the ward nurse did not know the type of mixed drug preparation injected by the patient.

ELIGIBILITY:
Inclusion Criteria:

1. age in the range of 50 to 85 years old
2. patients with knee osteoarthritis requiring primary unilateral total knee replacement
3. the body mass index in the range of 18 to 36 kg/m2
4. possess the physical status I-III of American Society of Anesthesiologists
5. the patient and his family members agree and sign the informed consent

Exclusion Criteria:

1. Non-osteoarthritis (rheumatoid arthritis, traumatic arthritis, septicemic arthritis, etc.)
2. History of knee surgery or knee injury, such as high tibial osteotomy, meniscus repair, ligament reconstruction, etc
3. Flexion deformity ≥30°, internal and external varus deformity ≥15°
4. People allergic to the drugs used in this study
5. Patients who had used glucocorticoids within 3 months before surgery

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
pain visual analogue scale score | 2 hours after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 4 hours after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 8 hours after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 24 hours after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 48 hours after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 72 hours after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 2 weeks after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 4 weeks after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 8 weeks after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect
pain visual analogue scale score | 12 weeks after surgery
  pain visual analogue scale score; range from 0 to 10; The lower it is, the better the analgesic effect

SECONDARY OUTCOMES:
Blood routine | Postoperative day 1
  Assay index including white blood cell count and neutrophil count.
Blood routine | Postoperative day 2
  Assay index including white blood cell count and neutrophil count.
Blood routine | Postoperative day 3
  Assay index including white blood cell count and neutrophil count.
Test index of drainage liquefaction | Postoperative day 1
  Assay index
Complication rate | Three months after surgery
  Follow-up visit
The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index | Three months after surgery
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index; range from 0 to 100; A higher score indicates better knee function
Knee range of motion | Postoperative day 1
  The rehabilitation doctor takes the measurements of changes in knee joint motion during the first three days after surgery
Knee range of motion | Postoperative day 2
  The rehabilitation doctor takes the measurements of changes in knee joint motion during the first three days after surgery
Knee range of motion | Postoperative day 3
  The rehabilitation doctor takes the measurements of changes in knee joint motion during the first three days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tian Hua, doctor, Study Chair — Director
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided